CLINICAL TRIAL: NCT02474966
Title: Effects of Deep Transcranial Magnetic Stimulation on the Permeability of the Blood-brain Barrier in Patients With Glioblastoma Multiforme: a Pilot Study
Brief Title: Effect of Deep TMS on the Permeability of the BBB in Patients With Glioblastoma Multiforme: a Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Maurizio Inghilleri, Principal Investigator, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 3403/23.10.14
Record Dates: First submitted 2015-06-11; First posted 2015-06-18 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Glioblastoma Multiforme of Brain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Real-Sham dTMS (Experimental): This arm will be treated before with real deep Transcranial Magnetic Stimulation (dTMS) (the first day) and after with sham dTMS (the second day)
  Interventions: Device: Deep Transcranial Magnetic Stimulation (dTMS)
- Sham-Real dTMS (Experimental): This arm will be treated before with sham deep Transcranial Magnetic Stimulation (dTMS) (the first day) and after with real dTMS (the second day)
  Interventions: Device: Deep Transcranial Magnetic Stimulation (dTMS)

INTERVENTIONS:
Device: Deep Transcranial Magnetic Stimulation (dTMS) — Patients will present on two consecutive days in order to receive dTMS followed by dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI). Subjects will be randomized into two groups: the first group will be treated before with real-dTMS (the first day) and after with sham-dTMS (the second day); the second group will be treated before with sham-dTMS (the first day) and after with realTMS (the second day). At the end of each session of dTMS the patients will undergo by MRI exams.

SUMMARY:
The blood-brain barrier (BBB) is a specialized interface allowing a unique environment for neuro-glia networks. BBB dysfunction is common in brain disorders. The Transcranial Magnetic Stimulation (TMS) is a non-invasive method of stimulating cortical motor neurons with the use of rapidly changing electromagnetic fields generated by a coil placed over the scalp. The objective of this study is to evaluate the safety and effects of the deep TMS (dTMS) on barrier integrity in patients with malignant glial tumors. BBB permeability will be quantified using dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI). Permeability change will be compared between two DCE-MRI scans performed immediately after "real" and "sham" rTMS, randomly assigned within one week of each other.

DETAILED DESCRIPTION:
The blood-brain barrier (BBB) is a specialized interface allowing a unique environment for neuro-glia networks. BBB dysfunction is common in brain disorders. However, the mechanisms underlying BBB opening are poorly understood. The investigators suggest a novel mechanism modulating BBB integrity and therapeutic implications in patients with glioblastoma multiforme. The Transcranial Magnetic Stimulation (TMS) is a noninvasive method of stimulating cortical motor neurons through the scalp and skull capable of inducing electrical currents and depolarizing neurons in focal brain areas with the use of rapidly changing electromagnetic fields generated by a coil placed over the scalp. The objective of this study is to evaluate the safety and effects of the deep TMS (dTMS) on barrier integrity in 20 patients with malignant glial tumors (glioblastoma multiforme). BBB permeability will be quantified using dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI). Permeability change will be compared between two DCE-MRI scans performed immediately after "real" and "sham" dTMS, randomly assigned within one week of each other.

Design of study: Randomized double-blind crossover study. Patients will present on two consecutive days in order to receive dTMS followed by DCE-MRI. Subjects will be randomized into two groups: the first group will be treated before with real-dTMS (the first day) and after with sham-dTMS (the second day); the second group will be treated before with sham-dTMS (the first day) and after with real-dTMS (the second day). At the end of each session of dTMS the patients will undergo by MRI exams.

Enrolled patients: twenty patients with glioblastoma multiforme treated with craniotomy and gross tumor resection or maximal debulking at least a year prior to the study and treated with standard post-operative radiotherapy and adjuvant chemotherapy.

dTMS will be delivered at 1 Hz, on the anterior periphery of the resected tumor bed using the Hesed-coil (H-coil) (Brainsway Ltd., Jerusalem, Israel). Sham stimulation will be delivered with a sham coil placed in the same helmet able to produce similar sounds and scalp sensations.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of glioblastoma multiforme (WHO grade IV)
* Craniotomy with resection of the tumor at least one year prior to the study
* Treatment with steroids or chemotherapy stable for at least four weeks prior to study enrollment

Exclusion Criteria:

* History of epilepsy
* Presence of cardiac pacemaker
* Presence of neurostimulators
* Presence of surgical clips or medical pumps
* Allergy to contrast medium for Magnetic Resonance Imaging
* History of head injuries
* Alcoholism or drugs abuse
* State of pregnant or breastfeeding
* Severe psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in blood-brain barrier permeability | Six months
  The efficacy of the deep Transcranial Magnetic Stimulation (dTMS) in modulating blood-brain barrier permeability in patients with glioblastoma multiforme through the measurement of the average value of the slope-value distribution function (CDF) evidenced with dynamic contrast-enhanced magnetic resonance imaging

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | Six months
  To evaluate the safety of the deep Transcranial Magnetic Stimulation (dTMS) applied in patients with glioblastoma multiforme

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Inghilleri, Professor, Principal Investigator — University "Sapienza" of Rome

REFERENCES:
- [Result] Abbott NJ, Patabendige AA, Dolman DE, Yusof SR, Begley DJ. Structure and function of the blood-brain barrier. Neurobiol Dis. 2010 Jan;37(1):13-25. doi: 10.1016/j.nbd.2009.07.030. Epub 2009 Aug 5. PMID 19664713
- [Result] Bolwig TG, Hertz MM, Paulson OB, Spotoft H, Rafaelsen OJ. The permeability of the blood-brain barrier during electrically induced seizures in man. Eur J Clin Invest. 1977 Apr;7(2):87-93. doi: 10.1111/j.1365-2362.1977.tb01578.x. PMID 404164
- [Result] Cote J, Bovenzi V, Savard M, Dubuc C, Fortier A, Neugebauer W, Tremblay L, Muller-Esterl W, Tsanaclis AM, Lepage M, Fortin D, Gobeil F Jr. Induction of selective blood-tumor barrier permeability and macromolecular transport by a biostable kinin B1 receptor agonist in a glioma rat model. PLoS One. 2012;7(5):e37485. doi: 10.1371/journal.pone.0037485. Epub 2012 May 21. PMID 22629405
- [Result] Hirschberg H, Uzal FA, Chighvinadze D, Zhang MJ, Peng Q, Madsen SJ. Disruption of the blood-brain barrier following ALA-mediated photodynamic therapy. Lasers Surg Med. 2008 Oct;40(8):535-42. doi: 10.1002/lsm.20670. PMID 18798293
- [Result] Pardridge WM. The blood-brain barrier: bottleneck in brain drug development. NeuroRx. 2005 Jan;2(1):3-14. doi: 10.1602/neurorx.2.1.3. PMID 15717053
- [Result] Prager O, Chassidim Y, Klein C, Levi H, Shelef I, Friedman A. Dynamic in vivo imaging of cerebral blood flow and blood-brain barrier permeability. Neuroimage. 2010 Jan 1;49(1):337-44. doi: 10.1016/j.neuroimage.2009.08.009. Epub 2009 Aug 12. PMID 19682584
- [Result] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Result] Roth Y, Zangen A, Hallett M. A coil design for transcranial magnetic stimulation of deep brain regions. J Clin Neurophysiol. 2002 Aug;19(4):361-70. doi: 10.1097/00004691-200208000-00008. PMID 12436090
- [Result] Wassermann EM, Zimmermann T. Transcranial magnetic brain stimulation: therapeutic promises and scientific gaps. Pharmacol Ther. 2012 Jan;133(1):98-107. doi: 10.1016/j.pharmthera.2011.09.003. Epub 2011 Sep 7. PMID 21924290
- [Result] Zangen A, Roth Y, Voller B, Hallett M. Transcranial magnetic stimulation of deep brain regions: evidence for efficacy of the H-coil. Clin Neurophysiol. 2005 Apr;116(4):775-9. doi: 10.1016/j.clinph.2004.11.008. Epub 2004 Dec 16. PMID 15792886
- [Result] Zimmermann R, Schmitt H, Rotter A, Sperling W, Kornhuber J, Lewczuk P. Transient increase of plasma concentrations of amyloid beta peptides after electroconvulsive therapy. Brain Stimul. 2012 Jan;5(1):25-9. doi: 10.1016/j.brs.2011.01.007. Epub 2011 Mar 12. PMID 22037136
- [Result] Sharp CD, Hines I, Houghton J, Warren A, Jackson TH 4th, Jawahar A, Nanda A, Elrod JW, Long A, Chi A, Minagar A, Alexander JS. Glutamate causes a loss in human cerebral endothelial barrier integrity through activation of NMDA receptor. Am J Physiol Heart Circ Physiol. 2003 Dec;285(6):H2592-8. doi: 10.1152/ajpheart.00520.2003. Epub 2003 Jul 31. PMID 12893641
- [Result] Mottaghy FM, Gangitano M, Horkan C, Chen Y, Pascual-Leone A, Schlaug G. Repetitive TMS temporarily alters brain diffusion. Neurology. 2003 May 13;60(9):1539-41. doi: 10.1212/01.wnl.0000058903.15205.46. PMID 12743250
- [Result] Chassidim Y, Veksler R, Lublinsky S, Pell GS, Friedman A, Shelef I. Quantitative imaging assessment of blood-brain barrier permeability in humans. Fluids Barriers CNS. 2013 Feb 7;10(1):9. doi: 10.1186/2045-8118-10-9. PMID 23388348
- [Result] Baker GJ, Yadav VN, Motsch S, Koschmann C, Calinescu AA, Mineharu Y, Camelo-Piragua SI, Orringer D, Bannykh S, Nichols WS, deCarvalho AC, Mikkelsen T, Castro MG, Lowenstein PR. Mechanisms of glioma formation: iterative perivascular glioma growth and invasion leads to tumor progression, VEGF-independent vascularization, and resistance to antiangiogenic therapy. Neoplasia. 2014 Jul;16(7):543-61. doi: 10.1016/j.neo.2014.06.003. PMID 25117977